CLINICAL TRIAL: NCT05643053
Title: Impact of Endotracheal Tube Fixation Methods on Tube Displacement During Pron Position
Brief Title: Comparison of Endotracheal Tube Fixation Methods in Prone Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Funda Atar, Diskapi Yildirim Beyazit Education and Research Hospital, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18/07/2022 142/05
Record Dates: First submitted 2022-11-23; First posted 2022-12-08 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Fixation Device; Complications
Keywords: endotracheal tube fixation; fiberoptic bronchoscopy; prone position

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- thomas fixation (Experimental)
  Interventions: Other: thomas fixation
- elastic band (Experimental)
  Interventions: Other: elastic band
- normal fixation adhesive tape (Experimental)
  Interventions: Other: normal fixation adhesive tape
- reinforced adhesive tape fixation (Experimental)
  Interventions: Other: reinforced adhesive tape fixation

INTERVENTIONS:
Other: thomas fixation — Use of the thomas tube holder for endotracheal tube fixation in patients operated in the prone position
  Arms: thomas fixation
Other: elastic band — Use of the elastic band for endotracheal tube fixation in patients operated in the prone position
  Arms: elastic band
Other: normal fixation adhesive tape — Use of the adhesive tape for endotracheal tube fixation in patients operated in the prone position
  Arms: normal fixation adhesive tape
Other: reinforced adhesive tape fixation — Use of the reinforced adhesive tape fixation for endotracheal tube fixation in patients operated in the prone position
  Arms: reinforced adhesive tape fixation

SUMMARY:
In particular, prone position surgeries risk potentially life-threatening ET tube dislocation. Failure to place the plaster used for ET tube fixation correctly and adequately in this position may contaminate the patch with body fluids and loosen the weight of the breathing circuit, causing the ET tube to slip and dislodge. Adhesive tape (plaster), bandage (non-adhesive), suturing, or a commercially available tube holding device are recommended for ET tube fixation in patients operated in the prone position. In addition, the adhesive plasters used can be taped on the patient's face to the maxilla, mandible, or both. Because of the urgent and critical settings, a fast, reliable, and easy-to-use method of ET tube fixation is invaluable as it will provide clinicians with greater confidence in the stability of alternative airways and reduce complications from airway maintenance. In our clinic, different fixation methods are used according to the experience and preference of the anesthesiologist. Our study aims to compare other fixation methods using FOB to fix the position of the ET tube with an appropriate method in prone position procedures and ensure that patients have safe airway management throughout the surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status I-II
* Mallampati score I-II

Exclusion Criteria:

* Patients who did not want to participate in the study
* Restricted mouth opening
* BMI ≥ 35 kg/m2
* Risk of airway malformation and aspiration (gastroesophageal reflux, hiatal -hernia, history of previous gastric surgery, GIS motility disorder)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-09 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Correct placement and subsequent fixation of the endotracheal tube in the prone patient | periopeative

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medical Science, Yıldırım Beyazıt Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh G, Manikandan S, Neema PK. Endotracheal tube fixation in neurosurgical procedures operated in prone position. J Anaesthesiol Clin Pharmacol. 2011 Oct;27(4):574-5. doi: 10.4103/0970-9185.86621. No abstract available. PMID 22096310